CLINICAL TRIAL: NCT05532683
Title: Development and Feasibility of a Lifestyle Group Intervention for Youth at Clinical High Risk for Psychosis
Brief Title: Feasibility Trial of a Lifestyle Intervention for CHR-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Bernalyn Ruiz-Yu, PhD, Postdoctoral Fellow, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB#22-001116
Record Dates: First submitted 2022-08-01; First posted 2022-09-08 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Prodromal Schizophrenia; Psychosis; Psychological Disorder; Psychological Stress
Keywords: early intervention; lifestyle intervention; clinical high risk for psychosis; health behavior
MeSH Terms: conditions — Schizotypal Personality Disorder; Psychotic Disorders; Mental Disorders; Stress, Psychological; Health Behavior

STUDY DESIGN:
Intervention Model Description: One group of 12 participants identified as at clinical high-risk for psychosis (CHR-P) will be recruited to participate in a 9-week health behavior promotion/lifestyle intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Behavior Group (Experimental): 9- week health behavior promotion group intervention
  Interventions: Behavioral: Health Behaviors Group

INTERVENTIONS:
Behavioral: Health Behaviors Group — The proposed intervention will include eight modules across nine weekly group sessions targeting psychoeducation of CHR-P symptoms, goal setting, physical activity, sleep, substance use, nutrition, and evidence-based strategies for stress management. Intervention facilitators will utilize motivational interviewing (MI; Miller & Rollnick, 2012) strategies to engage youth in goal setting to target change in health promotion behaviors. Caregivers will be invited to join at the end of each session for a 10-minute check-out where an outline of content covered and patient goals for the week will be shared.

SUMMARY:
The present study will assess the feasibility and social validity of an adjunctive health promotion group for youth and clinical high risk for psychosis (CHR-P). Youth participating in treatment at the Center for the Assessment and Prevention of Prodromal Sates (CAPPS) will be invited to participate in a weekly, adjunctive, closed psychoeducation group focused on sharing health promotion strategies and increasing health behaviors (e.g. improved sleep habits, increased participation in physical activity).

The aim of the group will be to provide psychoeducation on lifestyle risk and protective factors for youth at risk for psychosis (i.e. experiencing subthreshold psychosis symptoms). Topics covered will include psychoeducation, goal setting, stress management, sleep, physical activity, substance use, and nutrition. Evidence-based strategies to decrease risk factors and promote protective lifestyle factors for mental illness will be reviewed. Group leaders will utilize a motivational interviewing approach to facilitate the group.

The group will complete nine weekly group sessions. The goal of our research is to 1) determine the feasibility of a novel group-based health promotion intervention, 2) assess the social validity of the group, 3) measure the effects of the intervention on stress, sleep, physical activity, substance use, and nutrition, and 4) measure preliminary effects on symptoms and functioning.

ELIGIBILITY:
Inclusion Criteria:

1. between 13 and 17 years old
2. able to sign and provide informed consent (assent for minors)
3. meet criteria for CHR-P using the Structured Interview for Psychosis-Risk Syndromes (SIPS).
4. Must have a primary caregiver willing to participate who speaks fluent English

Exclusion Criteria:

1. current or lifetime DSM-5 psychotic disorder
2. impaired intellectual functioning (IQ <65)
3. history of neurological disorder
4. traumatic brain injury (≥7 on TBI screening tool)
5. significant substance use that makes CHR-P diagnosis ambiguous

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Participant Recruitment and Retention | Across Intervention: 9 weeks
  Feasibility will be measured by recruitment (participants approached/ participants enrolled) and retention (participants enrolled/ participants completed at least two-thirds of the intervention). Feasibility data will be summarized by the percent recruited, the percent retained by group and the mean and median number of sessions attended by group. The percent who attended each session by group over time will also be reported. Good feasibility will be defined as 70% of those enrolled completing at least two-thirds of the intervention (6 sessions).
Change in Physical Activity | Change from baseline (pre-intervention) to 9- week post-intervention
  The mean profile from baseline to post-treatment for physical activity as assessed by the International Physical Activity Questionnaire - Short Form (IPAQ-SF; Craig et al., 2017). Activity levels will be self-report.
Change Sleep Habits | Change from baseline (pre-intervention) to 9- week post-intervention
  Sleep will be assessed via self-report on the PROMIS Pediatric Sleep Disturbance scale (Buysse, et al., 2010). The Pediatric Sleep Disturbance Scale consists of 15 items rated 1 = Never, 2 = Almost Never, 3 = Sometimes, 4 = Almost Always, and 5 = Always, with a higher score indicating more sleep disturbance.
Change in Subjective Stress | Change from baseline (pre-intervention) to 9- week post-intervention
  Participant subjective stress will be assessed via the 10-item self-report Perceived Stress Scale ( PSS; Cohen et al., 1983).The PSS consists of 10 items rated 0= Never to 4= Very Often, with a higher score suggesting more stress.
Change in Substance Use | Change from baseline (pre-intervention) to 9- week post-intervention
  Alcohol and drug use will be measured by clinician rated on the Alcohol Use Scale and Drug Use Scale (AUS/DUS; Drake et al., 1996). This measure rates frequency and impairment associated with alcohol and drug use. Alcohol and drug use are rated on both frequency (0= no use to 5= almost daily) and impairment (0= abstinent to 5= dependence with institutionalization). A rating of 3 or higher on impairment corresponds with substance use disorder.
Change in Diet | Change from baseline (pre-intervention) to 9- week post-intervention
  Change in diet will be measured on the ASA24. This dietary assessment uses 24-hour recall to assess nutrition quality and provides measure of total energy intake and macronutrients.

SECONDARY OUTCOMES:
Social Validity as assessed by the Semi-Structured Interview for Social Validation | 9-week post-intervention
  The social validity of the intervention will be described qualitatively using a modified version of the Semi-Structured Interview for Social Validation. This interview measure includes questions directed at assessing the significance of the goals of the intervention, the acceptability of the procedures used, and the importance of the effects of the intervention. A thematic analysis procedure will be utilized for qualitative analysis of the interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). Treatment manual will also be made available. Proposals should be directed to bernalynruiz@mednet.ucla.edu. To gain access, data requestors will need to sign a data access agreement and provide methodologically sound research proposal.
Time Frame: Data will be made available beginning 3 months and ending 5 years following article publication.
Access Criteria: Those requesting access should have Ph.D. or equivalent level degree in psychology or a related field. Researchers should also provide a methodologically sound proposal.